CLINICAL TRIAL: NCT06987812
Title: Turkish Adaptation of The Mindful Eating Scale (MIND-EAT Scale): Validity and Reliability Study
Brief Title: Turkish Adaptation of the MIND-EAT Scale
Status: Recruiting | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Sponsor
Other Study IDs: Sedef Gungor-MIND-EAT scale-01
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Mindful Eating
Keywords: mindful eating, mindfulness, MIND-EAT, nutrition, Turkish scale

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Mindful eating is an important concept that refers to individuals regulating their eating behaviors by being aware of factors such as physical hunger, satiety, emotional states and environmental influences. This approach can be used especially in psychologically based interventions such as eating disorders, emotional eating and combating obesity.

Aim: In this study, it is aimed to adapt the MIND-EAT scale into Turkish and to analyze its validity and reliability.

Methods The sample of the study consists of at least 360 volunteer individuals aged 18 and over. Care will be taken to ensure a balanced gender distribution in the sample selection. The data collection process will be carried out through an online survey platform using non-probability random sampling method. In addition to obtaining information on the demographic characteristics (age, gender, education level, etc.) and eating habits of the participants through the survey, the Mindful Eating Scale (MIND-EAT Scale) will be applied as the main data collection tool. The Intuitive Eating Scale 2 (IES-2) and the Three Factor Eating Scale (TFEQ-R21) will be used to test the validity of the scale. To assess the reliability of the scale, a minimum of 20 participants will be administered the scale again at a 2-week interval.

Expected Results of the Study: If the MIND-EAT scale is adapted to the Turkish population with a validity and reliability study, it will determine whether individuals have eating awareness and will contribute to the development of more effective approaches.

DETAILED DESCRIPTION:
Although eating behavior is primarily a physiological response to hunger, social and cultural factors can also trigger eating even when there is no need to eat. Extrinsically motivated eating behavior cannot be regulated by the body's signals of satiety. Therefore, approaches such as mindful eating (ME) have been developed to reduce the influence of extrinsic motivation and increase the importance of intrinsic motivation and the sensory properties of food. ME is the state of focusing on and being mindful of food while eating. Although the goal is not weight loss, it is thought that paying attention to the experience of food can increase awareness of the impact of food on a person and lead to healthier choices. Mindfulness has proven positive effects on overall health and is recommended by the American Heart Association. Furthermore, mindfulness-based approaches have been shown to have positive effects on changing maladaptive eating behaviors in individuals of different weights. Given these positive aspects, it is important to have a comprehensive scale that covers all aspects of mindful eating and offers an overall scoring.

In this study, it is aimed to adapt the MIND-EAT scale into Turkish and to analyze its validity and reliability.

Type, Population and Sample of the Study:

The sample of the study will consist of individuals aged 18 and over. Individuals who are volunteers and have no communication problems will be included in the study. The approval of the participants will be obtained in the study, which will be started if the ethics committee approval is obtained. Care will be taken to ensure that the number of men and women in the sample is close to each other. In the validity and reliability study, data will be collected with an online questionnaire. In the internal construct validity phase of the study, it was aimed to reach at least 360 individuals by including at least 15 people for each item in the scale (24 x 15 = 360) for the sample size calculation.

The scale will be administered to at least 360 individuals aged 18 years and over by non-probability, random sampling method. A "participant number" will be given to the form filled out by each participant. The scale will be reapplied 2 weeks later to a minimum of 20 participants, which is required for test-retest reliability.

In this study, written permission was obtained by the developers of the MIND-EAT Scale via e-mail for the Turkish validity and reliability of the scale. Following the ethics committee permission, the language adaptation process of the MIND-EAT scale will be carried out first. The next stage will be the validity and reliability testing of the scale by applying it in the targeted sample.

Language Adaptation of the Scale:

For the language adaptation study of the original French language scale, the original scale will be independently translated into Turkish by three experts who are fluent in French. In language adaptation, standard translation-back translation method will be used to minimize expression differences. The process of adaptation of the scale into Turkish will be completed after the form obtained as a result of back-translation and the original version are evaluated in terms of consistency and semantic integrity by applying expert opinion and making the necessary arrangements.

Evaluation of the Linguistic Equivalence of the Scale:

In order to evaluate the linguistic equivalence of the finalized scale, at least 10 people who have the same characteristics as the study group and who have an advanced knowledge of French will be asked to apply the French and Turkish forms of the scale at 2-week intervals. The similarities between the applications of the scale in two languages will be examined and its linguistic validity will be evaluated.

Testing the Reliability of the Scale:

The finalized Turkish scale will be administered to a sample of at least 360 participants. The consistency of the responses to the scale items will be examined with Cronbach alpha coefficient. The item-total correlation coefficient will also be calculated for each item. In the evaluation of test-retest reliability, it is planned to reapply the scale to at least 20 participants with an interval of 2 weeks.

Testing the Validity of the Scale:

Intuitive Eating Scale 2 (IES-2) and Three Factor Eating Scale (TFEQ-R21) will be used to test the criterion-related validity of the MIND-EAT Scale. It was decided to apply the Intuitive Eating Scale 2 and the Trifactor Eating Scale to the study sample in the evaluation of the relationship between these two scales, which were predicted to show an above average relationship with the scale whose validity was evaluated The reason for selecting the Intuitive Eating Scale 2 and the Trifactor Eating Scales for testing the criterion-related validity; Both intuitive eating and eating mindfulness enable individuals to encourage conscious regulation of their eating behaviors, while eating mindfulness, as measured in the Three-factor eating scale, can help balance behaviors such as emotional and external eating and help one develop a healthier eating pattern based on internal signals. When used together, these scales can contribute to individuals' deeper understanding and control of their eating behaviors. The construct validity of the MIND-EAT scale is assessed by exploratory and confirmatory factor analysis.

Data Collection Tools:

General information of the participants:

General characteristics of the participants such as age, gender, weight, height, education, disease status and information about their eating habits will be recorded.

MIND-EAT scale:

This scale was developed by Van Beekum et al. as a comprehensive measure of mindful eating behaviors in which responses are rated on a 5-point frequency scale ranging from 1 "never or almost never" to 5 "always or almost always". It consists of 6 sub-dimensions and includes 24 items. The scale score is obtained by dividing the score obtained from the items by the number of items. Sub-dimension scores can also be calculated by dividing the score obtained from the questions related to each sub-dimension by the number of questions in the sub-dimension. The scale has no cut-off point. For the Turkish validity and reliability of the scale, written permission was obtained from Van Beekum via e-mail.

Intuitive Eating Scale 2 (IES-2):

The Intuitive Eating Scale (IES) is a 21-item scale developed by Tylka and colleagues in 2006 to measure intuitive eating behavior. Later, an improved version of the scale, the Intuitive Eating Scale-2 (IES-2), was created by Tylka and Kroon Van Diest in 2013. The IES-2 has a 23-item structure by adding 12 new items to the 11 items in the original scale. The IES-2, which has four subscales, assesses the following dimensions: eating for physical rather than emotional reasons; unconditional permission to eat; trust in hunger and satiety signals; and congruence of body-food choices. The Turkish adaptation of the scale was conducted by Bakıner and the internal consistency coefficient was found to be 0.89. It is accepted that the higher the score obtained from the scale, the higher the intuitive eating behavior of the individual.

Three Factor Eating Scale (TFEQ-R21):

The Three-Factor Eating Scale (TFEQ) developed by Stunkard and Messick is a tool used to measure eating behavior. This scale, which was adapted into Turkish by Karakuş et al. consists of 21 items and is named as TFEQ-R21. The scale is used to assess uncontrolled eating behavior and consists of three subscales. Uncontrolled eating is defined as the loss of control while eating without any external factor or feeling of hunger.

Data Collection:

Data will be collected by the researchers. Expected Results of the Study: If the MIND-EAT scale is adapted to the Turkish population with a validity and reliability study, it will determine whether individuals have eating awareness and will contribute to the development of more effective approaches.

ELIGIBILITY:
Inclusion criteria:

Individuals 18 years of age and older Volunteers, individuals with no communication problems will be included in the study.

Exclusion criteria:

Individuals under 18 years of age, Individuals with communication problems and Individuals with any psychological disorder will not be included in the study.

Min Age: 18 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population of this study consists of male and female individuals aged 18 years and over.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Testing scale reliability | Up to one month
  In the evaluation of test-retest reliability, it is planned to reapply the scale to at least 20 participants with an interval of 2 weeks.

SECONDARY OUTCOMES:
Testing the validity of the scale | Up to one month
  Testing the Validity of the ScaleIntuitive Eating Scale 2 (IES-2) and Three-Factor Eating Scale (TFEQ-R21) will be used to test the criterion-related validity of the MIND-EAT Scale. It was decided to apply the Intuitive Eating Scale 2 and the Three-Factor Eating Scale to the research sample in the evaluation of the relationship between these two scales, which were predicted to show an above average relationship with the scale whose validity was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Mathieu J. What should you know about mindful and intuitive eating? J Am Diet Assoc. 2009 Dec;109(12):1982-7. doi: 10.1016/j.jada.2009.10.023. No abstract available. PMID 19942013
- [Background] Grider HS, Douglas SM, Raynor HA. The Influence of Mindful Eating and/or Intuitive Eating Approaches on Dietary Intake: A Systematic Review. J Acad Nutr Diet. 2021 Apr;121(4):709-727.e1. doi: 10.1016/j.jand.2020.10.019. Epub 2020 Dec 3. PMID 33279464
- [Background] Tapper K. Mindful eating: what we know so far. Nutr Bull. 2022 Jun;47(2):168-185. doi: 10.1111/nbu.12559. Epub 2022 May 10. PMID 36045097
- [Background] Lee EKP, Yeung NCY, Xu Z, Zhang D, Yu CP, Wong SYS. Effect and Acceptability of Mindfulness-Based Stress Reduction Program on Patients With Elevated Blood Pressure or Hypertension: A Meta-Analysis of Randomized Controlled Trials. Hypertension. 2020 Dec;76(6):1992-2001. doi: 10.1161/HYPERTENSIONAHA.120.16160. Epub 2020 Nov 2. PMID 33131316
- [Background] Scott-Sheldon LAJ, Gathright EC, Donahue ML, Balletto B, Feulner MM, DeCosta J, Cruess DG, Wing RR, Carey MP, Salmoirago-Blotcher E. Mindfulness-Based Interventions for Adults with Cardiovascular Disease: A Systematic Review and Meta-Analysis. Ann Behav Med. 2020 Jan 1;54(1):67-73. doi: 10.1093/abm/kaz020. PMID 31167026
- [Background] Levine GN, Cohen BE, Commodore-Mensah Y, Fleury J, Huffman JC, Khalid U, Labarthe DR, Lavretsky H, Michos ED, Spatz ES, Kubzansky LD. Psychological Health, Well-Being, and the Mind-Heart-Body Connection: A Scientific Statement From the American Heart Association. Circulation. 2021 Mar 9;143(10):e763-e783. doi: 10.1161/CIR.0000000000000947. Epub 2021 Jan 25. PMID 33486973
- [Background] Peitz D, Schulze J, Warschburger P. Getting a deeper understanding of mindfulness in the context of eating behavior: Development and validation of the Mindful Eating Inventory. Appetite. 2021 Apr 1;159:105039. doi: 10.1016/j.appet.2020.105039. Epub 2020 Nov 10. PMID 33186622
- [Background] Osborne JW. & Costello AB. Sample size and subject to item ratio in principal components analysis. Pract Assess Res & Eval, 2004;9:1-9.
- [Background] Sperber AD. Translation and validation of study instruments for cross-cultural research. Gastroenterology. 2004 Jan;126(1 Suppl 1):S124-8. doi: 10.1053/j.gastro.2003.10.016. PMID 14978648
- [Background] Akırmak, Ü., Bakıner, E., Bolak Boratav, H. & Güneri, G. Cross-cultural adaptation of the intuitive eating scale-2: psychometric evaluation in a sample in Turkey. Current Psychology, 2018; 40: 1083-1093.
- [Background] Karakuş, S. Ş., Yıldırım, H., & Büyüköztürk, Ş. Üç Faktörlü Yeme Ölçeğinin Türk kültürüne uyarlanması: Geçerlik ve güvenirlik çalışması. TAF Preventive Medicine Bulletin, 2016; 15(3): 229-237. DOI: 10.5455/pmb.1-1446540396.
- [Background] Van Beekum M, Shankland R, Rodhain A, Robert M, Marchand C, Herry A, Prioux C, Touvier M, Barday M, Turgon R, Avignon A, Leys C, Peneau S. Development and validation of the mindful eating scale (mind-eat scale) in a general population. Appetite. 2024 Aug 1;199:107398. doi: 10.1016/j.appet.2024.107398. Epub 2024 May 6. PMID 38710449
- [Background] Tylka TL, Kroon Van Diest AM. The Intuitive Eating Scale-2: item refinement and psychometric evaluation with college women and men. J Couns Psychol. 2013 Jan;60(1):137-53. doi: 10.1037/a0030893. PMID 23356469
- [Background] Bakıner, E. (2017). Turkish adaptation of the Intuitive Eating Scale-2. Yüksek Lisans Tezi. İstanbul Bilgi Üniversitesi, İstanbul.
- [Background] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480